CLINICAL TRIAL: NCT07093034
Title: Sustained Auricular Nerve Stimulation for PVC Suppression
Acronym: SANS-PVC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Parasym Ltd. (Industry); Zywie Healthcare (Unknown)
Responsible Party: Principal Investigator, Ulrika Birgersdotter-Green, Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 812185
Record Dates: First submitted 2025-07-14; First posted 2025-07-30 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-08

CONDITIONS: Premature Ventricular Complexes; PVC - Premature Ventricular Contraction; Auricular Vagus Nerve Stimulation
Keywords: auricular vagus nerve stimulation; parasym; premature ventricular contractions (PVCs); Non-invasive neuromodulation; Cardiac arrhythmia; autonomic nervous system modulation; Trancutaneous electrical stimulation; Randomized controlled trial; heart rate variability; feasibility study
MeSH Terms: conditions — Ventricular Premature Complexes; Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Arm 1: Active stimulation followed by crossover to Sham stimulation (Experimental)
  Interventions: Device: Extended nocturnal use of auricular vagus nerve stimulator device
- Arm 2: Sham stimulation followed by crossover to Active stimulation (Experimental)
  Interventions: Device: Extended nocturnal use of auricular vagus nerve stimulator device

INTERVENTIONS:
Device: Extended nocturnal use of auricular vagus nerve stimulator device — Patients will wear the ParasymTM device with an ear clip on the tragus that provides stimulation at sub-detection threshold.

SUMMARY:
Non-invasive vagus nerve stimulation has been clinically tested for the treatment cardiac arrhythmias. However, prior studies have shown mixed results-possibly in part due to inadequate stimulation duration. Therefore, we have designed an investigator-initiated early feasibility study to evaluate safety, tolerability, and compliance with prolonged, nocturnal auricular nerve stimulation using the Parasym device.

DETAILED DESCRIPTION:
The study will utilize the Parasym transcutaneous auricular vagal nerve stimulation device. This small, battery-powered device delivers electrical stimulation through an ear clip attached to the tragus. Participants will self-administer the stimulation once daily, at bedtime, for 6 continuous hours. The device has two settings to facilitate our RCT: active treatment and sham control. After one month in the first treatment arm, participants will be crossed over to the other arm of the study. Participants and outcome assessors will be blinded to the allocation. The primary outcomes will be assessed via standardized questionnaires administered by blinded outcome assessors. The secondary outcome of PVC burden will be assessed by non-invasive event monitors.

ELIGIBILITY:
Inclusion Criteria

Individuals must meet all of the following inclusion criteria to be eligible to participate in this study:

Age ≥ 18 years

PVC burden ≥ 5% documented on an event monitor or implanted cardiac device

Provide written informed consent

Willingness to comply with all study procedures

Availability for the duration of the study (10 weeks)

Individuals meeting any of the following exclusion criteria at baseline will be excluded from study participation:

Unwilling or unable to provide informed consent for oneself

Last available left ventricular ejection fraction < 20%

NYHA Class IV symptoms

Acute coronary syndrome within two weeks of randomization

Active pregnancy or breastfeeding

Intention to become pregnant

Statement Regarding Equitable Selection:

This study will not exclude specific populations based on age, sex, race, or ethnicity. The inclusion/exclusion criteria are based on clinical factors relevant to the study intervention and the safety of participants. Limited English proficiency will not be an exclusion criterion, and appropriate translation services will be provided to ensure informed consent and understanding of study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Safety | 10 weeks (duration of entire study)
  The occurrence of adverse events (AEs) throughout the study.
Tolerability | 10 weeks
  Participants will rate tolerability of wearing the device at night at multiple pre-specified time points throughout the study
Quality of Life | 10 weeks
  Participants will rate quality of life at multiple pre-specified time points throughout the study
Feasibility | 10 weeks
  Participants will rate ease of wearing the device at night at multiple pre-specified time points throughout the study

SECONDARY OUTCOMES:
PVC burden | 10 weeks
  PVC burden will be tracked by event monitoring at pre-specified time points throughout the study

OTHER OUTCOMES:
PVC Burden stratified by timing | 10 weeks
  PVC burden during night time 12 hours and day time 12 hours will be compared to see if there is a significant difference
Heart rate variability (HRV) | 10 weeks
  HRV will be tracked throughout the study via event monitors at prespecified time points

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego Health System, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared if requested by the receiving journal or reviewer. We will de-identify the data prior to providing this information.

REFERENCES:
- [Result] Kim AY, Marduy A, de Melo PS, Gianlorenco AC, Kim CK, Choi H, Song JJ, Fregni F. Safety of transcutaneous auricular vagus nerve stimulation (taVNS): a systematic review and meta-analysis. Sci Rep. 2022 Dec 21;12(1):22055. doi: 10.1038/s41598-022-25864-1. PMID 36543841
- [Result] Gentile F, Giannoni A, Navari A, Degl'Innocenti E, Emdin M, Passino C. Acute right-sided transcutaneous vagus nerve stimulation improves cardio-vagal baroreflex gain in patients with chronic heart failure. Clin Auton Res. 2025 Feb;35(1):75-85. doi: 10.1007/s10286-024-01074-9. Epub 2024 Oct 14. PMID 39402309
- [Result] Hua K, Cummings M, Bernatik M, Brinkhaus B, Usichenko T, Dietzel J. Cardiovascular effects of auricular stimulation -a systematic review and meta-analysis of randomized controlled clinical trials. Front Neurosci. 2023 Sep 1;17:1227858. doi: 10.3389/fnins.2023.1227858. eCollection 2023. PMID 37727325
- [Result] Frangos E, Ellrich J, Komisaruk BR. Non-invasive Access to the Vagus Nerve Central Projections via Electrical Stimulation of the External Ear: fMRI Evidence in Humans. Brain Stimul. 2015 May-Jun;8(3):624-36. doi: 10.1016/j.brs.2014.11.018. Epub 2014 Dec 6. PMID 25573069
- [Result] Stavrakis S, Stoner JA, Humphrey MB, Morris L, Filiberti A, Reynolds JC, Elkholey K, Javed I, Twidale N, Riha P, Varahan S, Scherlag BJ, Jackman WM, Dasari TW, Po SS. TREAT AF (Transcutaneous Electrical Vagus Nerve Stimulation to Suppress Atrial Fibrillation): A Randomized Clinical Trial. JACC Clin Electrophysiol. 2020 Mar;6(3):282-291. doi: 10.1016/j.jacep.2019.11.008. Epub 2020 Jan 29. PMID 32192678
- [Result] Stavrakis S, Chakraborty P, Farhat K, Whyte S, Morris L, Abideen Asad ZU, Karfonta B, Anjum J, Matlock HG, Cai X, Yu X. Noninvasive Vagus Nerve Stimulation in Postural Tachycardia Syndrome: A Randomized Clinical Trial. JACC Clin Electrophysiol. 2024 Feb;10(2):346-355. doi: 10.1016/j.jacep.2023.10.015. Epub 2023 Nov 22. PMID 37999672
- [Result] Chakraborty P, Farhat K, Morris L, Whyte S, Yu X, Stavrakis S. Non-invasive Vagus Nerve Simulation in Postural Orthostatic Tachycardia Syndrome. Arrhythm Electrophysiol Rev. 2023 Dec 13;12:e31. doi: 10.15420/aer.2023.20. eCollection 2023. PMID 38173801
- [Result] Premchand RK, Sharma K, Mittal S, Monteiro R, Dixit S, Libbus I, DiCarlo LA, Ardell JL, Rector TS, Amurthur B, KenKnight BH, Anand IS. Autonomic regulation therapy via left or right cervical vagus nerve stimulation in patients with chronic heart failure: results of the ANTHEM-HF trial. J Card Fail. 2014 Nov;20(11):808-16. doi: 10.1016/j.cardfail.2014.08.009. Epub 2014 Sep 1. PMID 25187002
- [Result] Gold MR, Van Veldhuisen DJ, Hauptman PJ, Borggrefe M, Kubo SH, Lieberman RA, Milasinovic G, Berman BJ, Djordjevic S, Neelagaru S, Schwartz PJ, Starling RC, Mann DL. Vagus Nerve Stimulation for the Treatment of Heart Failure: The INOVATE-HF Trial. J Am Coll Cardiol. 2016 Jul 12;68(2):149-58. doi: 10.1016/j.jacc.2016.03.525. Epub 2016 Apr 4. PMID 27058909
- [Result] Zannad F, De Ferrari GM, Tuinenburg AE, Wright D, Brugada J, Butter C, Klein H, Stolen C, Meyer S, Stein KM, Ramuzat A, Schubert B, Daum D, Neuzil P, Botman C, Castel MA, D'Onofrio A, Solomon SD, Wold N, Ruble SB. Chronic vagal stimulation for the treatment of low ejection fraction heart failure: results of the NEural Cardiac TherApy foR Heart Failure (NECTAR-HF) randomized controlled trial. Eur Heart J. 2015 Feb 14;36(7):425-33. doi: 10.1093/eurheartj/ehu345. Epub 2014 Aug 31. PMID 25176942
- [Result] De Ferrari GM, Crijns HJ, Borggrefe M, Milasinovic G, Smid J, Zabel M, Gavazzi A, Sanzo A, Dennert R, Kuschyk J, Raspopovic S, Klein H, Swedberg K, Schwartz PJ; CardioFit Multicenter Trial Investigators. Chronic vagus nerve stimulation: a new and promising therapeutic approach for chronic heart failure. Eur Heart J. 2011 Apr;32(7):847-55. doi: 10.1093/eurheartj/ehq391. Epub 2010 Oct 28. PMID 21030409
- [Result] Li M, Zheng C, Sato T, Kawada T, Sugimachi M, Sunagawa K. Vagal nerve stimulation markedly improves long-term survival after chronic heart failure in rats. Circulation. 2004 Jan 6;109(1):120-4. doi: 10.1161/01.CIR.0000105721.71640.DA. Epub 2003 Dec 8. PMID 14662714
- [Result] Eckberg DL, Drabinsky M, Braunwald E. Defective cardiac parasympathetic control in patients with heart disease. N Engl J Med. 1971 Oct 14;285(16):877-83. doi: 10.1056/NEJM197110142851602. No abstract available. PMID 4398792